CLINICAL TRIAL: NCT04059627
Title: Feasibility of the "Heart-track" Rehabilitative Device Prototype Designed for Exercise Training Post Coronary Revascularisation
Brief Title: Feasibility of the "Heart-track" Rehabilitative Device Prototype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Eng Chan Neoh, Senior Physiotherapist, Tan Tock Seng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018/00307
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Cardiac Infarct; Cardiac Event
Keywords: Cardiac Rehab
MeSH Terms: conditions — Myocardial Infarction; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Twelve community-dwelling adults who are also active member of cardiac rehab support group, aged above 50, and undergone coronary revascularisation for acute myocardial infarction at least 1 year before were recruited.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Participants were introduced to "Heart-Track" mobile app system and its navigational characteristics with standardised instructions. Each participant then performed a self-directed Cardiac rehabilitation session using the app.
  Interventions: Device: Heart Track

INTERVENTIONS:
Device: Heart Track — Description of the device: Wearable heart rate sensors are used in Heart-track, and a receiver on a smartphone app. Real-time wireless heart rate data is sent to paired mobile device with a wireless distance of up to 10m. The sensor is able to monitor a heart rate range of 30 to 240 beats per minute.
  Another component of Heart-track is a "Heart-track" mobile app which captures and reflect real-time heart rate from the heart rate sensor. The mobile app also includes warm-up and cool down exercises that are gamified and supported on a smart-phone running on Android or iOS platforms.
  The HR sensor will be purchased by our collaborator, Immersive Play Pte Ltd.

SUMMARY:
Abstract Title: "Heart-track" cardiac rehabilitation device prototype designed for exercise training post coronary revascularisation: A usability study Background: Percutaneous Coronary Intervention (PCI) is a common surgical procedure for heart attack patients. International guidelines recommend that all patients complete phase two (outpatient) cardiac rehabilitation (CR) after PCI, as it plays a critical role in reducing five-year cardiovascular mortality and the risk of cardiovascular-related hospital admission. Patients in our institution have suboptimal exercise compliance and effectiveness during cardiac rehabilitation. Root cause analysis identified 'lack of commitment', 'lack of care monitoring and continuity' and 'lack of motivation and engagement' to be key contributing factors. Yet, healthcare resource limitations necessitate innovation for care continuity and patient engagement. "Heart-track", a novel, app-based innovation was created. By 'game-ifying' cardiac rehabilitative exercise training program, "Heart-track" guides and tracks cardiac rehabilitation at home at patient's comfort.

Purpose: To explore experiences of app usability in terms of content, functionality and design of the prototype "Heart-track" app to improve user experience.

Methods: Twelve community-dwelling adults who are also active member of cardiac rehab support group, aged above 50, and undergone coronary revascularisation for acute myocardial infarction at least 1 year before were recruited. Participants were introduced to "Heart-Track" mobile app system and its navigational characteristics with standardised instructions. Each participant then performed a self-directed Cardiac rehabilitation session using the app. Participants rated their experience with the hardware and software components of "Heart Track", and their acceptance of it as a cardiac rehabilitation tool. Descriptive analysis of quantitative responses were analysed using IBM SPSS software version 19.0 (Armonk, NY: IBM Corp).

DETAILED DESCRIPTION:
Abstract Title: "Heart-track" cardiac rehabilitation device prototype designed for exercise training post coronary revascularisation: A usability study Background: Percutaneous Coronary Intervention (PCI) is a common surgical procedure for heart attack patients. International guidelines recommend that all patients complete phase two (outpatient) cardiac rehabilitation (CR) after PCI, as it plays a critical role in reducing five-year cardiovascular mortality and the risk of cardiovascular-related hospital admission. Patients in our institution have suboptimal exercise compliance and effectiveness during cardiac rehabilitation. Root cause analysis identified 'lack of commitment', 'lack of care monitoring and continuity' and 'lack of motivation and engagement' to be key contributing factors. Yet, healthcare resource limitations necessitate innovation for care continuity and patient engagement. "Heart-track", a novel, app-based innovation was created. By 'game-ifying' cardiac rehabilitative exercise training program, "Heart-track" guides and tracks cardiac rehabilitation at home at patient's comfort.

Purpose: To explore experiences of app usability in terms of content, functionality and design of the prototype "Heart-track" app to improve user experience.

Methods: Twelve community-dwelling adults who are also active member of cardiac rehab support group, aged above 50, and undergone coronary revascularisation for acute myocardial infarction at least 1 year before were recruited. Participants were introduced to "Heart-Track" mobile app system and its navigational characteristics with standardised instructions. Each participant then performed a self-directed Cardiac rehabilitation session using the app. Participants rated their experience with the hardware and software components of "Heart Track", and their acceptance of it as a cardiac rehabilitation tool. Descriptive analysis of quantitative responses were analysed using IBM SPSS software version 19.0 (Armonk, NY: IBM Corp).

ELIGIBILITY:
Inclusion Criteria:

* Minimum 21 to 65 years of age
* conversational fluency in English
* undergone coronary revascularisation for acute myocardial infarction within last 5 years
* last documented ejection fraction of at least 40%
* completed a minimum of eight supervised CR sessions
* exercises at least once a week for a minimum duration of thirty minutes
* at least 6 months' experience using a smartphone
* recent experience(at least one months' experience) with any mobile app
* displaying capacity for self-monitoring and entering data.

Exclusion Criteria:

-Abnormal physiological response during exercise

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Survey | through study completion, an average of 3 months
  Participants rated their experience with the hardware and software components of "Heart Track", and their acceptance of it as a cardiac rehabilitation tool. The survey form is a likert-scale ( Strongly agree to strongly disagree) survey that asking subjects about their feedback and satisfaction about the Heart Track hardware and software, and overall experience using Heart Track.

CONTACTS AND LOCATIONS:
Overall Officials: Eng Chuan Neoh, masters, Study Director — Senior Physiotherapist
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No